CLINICAL TRIAL: NCT02828293
Title: Understanding GMK Sphere Implant Tibiofemoral Kinematics by Means of Dynamic Videofluoroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.014.11
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2017-09

CONDITIONS: Arthroplasty; Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- GMK Sphere: Patients who underwent total knee replacement using GMK Sphere implants. Patients underwent surgery before the inclusion in the study.
  Interventions: Other: Dynamic videofluoroscopic analysis
- GMK PS Fixed Bearing: Patients who underwent total knee replacement using GMK PS Fixed Bearing implants. Patients underwent surgery before the inclusion in the study.
  Interventions: Other: Dynamic videofluoroscopic analysis
- GMK UC Fixed Bearing: Patients who underwent total knee replacement using GMK UC Fixed Bearing implants. Patients underwent surgery before the inclusion in the study.
  Interventions: Other: Dynamic videofluoroscopic analysis

INTERVENTIONS:
Other: Dynamic videofluoroscopic analysis — Patients bearing 3 different prosthesis (3 groups) will be prospactively assessed with videofluoroscopy.

SUMMARY:
The objective of this research project is to perform a comparative study on the in vivo kinematics of the GMK Sphere prosthesis in comparison to the conventional GMK PS Fixed Bearing TKA and the GMK UC Fixed Bearing TKA.

ELIGIBILITY:
Inclusion Criteria:

* subjects bearing a TKA with one of the studied prosthesis
* male and female older than 18 years old
* patients who are willing and able to sign an informed consent form

Exclusion Criteria:

* any case not described in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 8-10 subjects with Medacta GMK Sphere TKA, 8-10 subjects with GMK PS Fixed Bearing TKA and 8-10 subjects with a GMK UC Fixed Bearing TKA will be involved in this project.
  The subject recruitment will be based on the clinical reports of the follow-up examination including the standard clinical assessed parameters alignment, the Western Ontario and McMaster Universities Arthritis Index (WOMAC) and the visual analog scale (VAS)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
2D/3D videofluoroscopy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomechanics ETH Zurich, Zurich, Switzerland